CLINICAL TRIAL: NCT01205217
Title: Randomized Study of Efficacy & Safety of Lapatinib & Epirubicin & Cyclophosphamide (EC90) Followed by Paclitaxel & Lapatinib Compared With EC90 Followed by Paclitaxel & Trastuzumab, as Neoadjuvant Therapy in Patients With Previously Untreated ErbB2-overexpressing Stage I - IIIA Breast Cancer.
Brief Title: Lapatinib or Trastuzumab Given Prior to Surgery With Chemotherapy in Patients With Early Breast Cancer
Acronym: ELATE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Data presented at SABCS 2010 showing that dual blockade is superior to monotherapy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113957
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; epirubicin; cyclophosphamide; trastuzumab; paclitaxel; neoadjuvant therapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; Trastuzumab; Epirubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Lapatinib in combination with epirubicin and cyclophosphamide followed by paclitaxel and lapatinib.
  Part I (Week 1-12) Epirubicin 90 mg/m2 by IV infusion on Day 1 every 21 days Cyclophosphamide 600 mg/m2 by IV infusion on Day 1 every 21 days Lapatinib 1000 mg orally once daily continuously Loperamide as required for the proactive management of diarrhoea
  Part II (Week 13-24) Paclitaxel 80 mg/m2 by IV infusion on Day 1 of each week Lapatinib 1000 mg orally once daily continuously Loperamide as required for the proactive management of diarrhoea
  Interventions: Drug: Lapatinib; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel
- Arm B (Active Comparator): Epirubicin and cyclophosphamide followed by paclitaxel and trastuzumab.
  Part I (Week 1-12) Epirubicin 90 mg/m2 by IV infusion on Day 1 every 21 days Cyclophosphamide 600 mg/m2 by IV infusion on Day 1 every 21 days
  Part II (Week 13-24) Paclitaxel 80 mg/m2 by IV infusion on Day 1 of each week Trastuzumab 4 mg/kg IV load followed by 2 mg/kg IV Day 1 of each week
  Interventions: Drug: Trastuzumab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Lapatinib — Lapatinib 1000 mg orally once daily continuously
  Arms: Arm A
Drug: Trastuzumab — Part II (Week 13-24) Trastuzumab 4 mg/kg IV load followed by 2 mg/kg IV Day 1 of each week
  Arms: Arm B
Drug: Epirubicin — Part I (Week 1-12) Epirubicin 90 mg/m2 by IV infusion on Day 1 every 21 days
Drug: Cyclophosphamide — Part I (Week 1-12) Cyclophosphamide 600 mg/m2 by IV infusion on Day 1 every 21 days
Drug: Paclitaxel — Part II (Week 13-24) Paclitaxel 80 mg/m2 by IV infusion on Day 1 of each week

SUMMARY:
This study will test the safety of a drug called lapatinib and how well it works. Lapatinib (also called Tyverb or Tykerb) will be compared with another drug trastuzumab (also called Herceptin).

Trastuzumab is an antibody against the HER2 protein. It binds to part of the HER2 protein to stop it working. Clinical trials have found that adding trastuzumab to chemotherapy lowers the rate of cancer recurrence and improves survival in women with HER2 positive breast cancer.

Lapatinib also stops the HER2 protein working and may slow or stop cancer cells from growing and may prevent cancer from returning. Lapatinib has been approved in some countries to treat patients with certain types of breast cancer. However lapatinib has not been approved to treat early breast cancer. This study is one of many being carried out involving lapatinib in early breast cancer and these studies are showing that it is a promising treatment.

This study will compare lapatinib and trastuzumab. One group of people will take lapatinib and another group will take trastuzumab. The effects of the drugs, both good and bad, will be compared. This study will compare two different durations of HER2 treatment to see if earlier introduction of HER2 treatment is beneficial. The lapatinib group will receive HER2 treatment from the very beginning for 24 weeks prior to surgery and the trastuzumab group will only receive HER2 therapy for 12 weeks prior to surgery.

DETAILED DESCRIPTION:
This is a randomized, parallel-arm, open-label, multicentre, Phase II study to determine the efficacy and safety of lapatinib in combination with epirubicin and cyclophosphamide (EC90-L) followed by paclitaxel and lapatinib (PX-L) compared with EC90 followed by paclitaxel and trastuzumab (PX-T) as systemic neoadjuvant therapy for patients with previously untreated, operable, ErbB2-overexpressing, Stage I- IIIA breast cancer.

Approximately 164 subjects will be enrolled in the study. Subjects will be randomised in a 1:1 ratio and stratified according to the following factors, each of which must be established prior to commencing randomisation:

* Tumour size (≤ 2 cm versus >2 cm in diameter).
* Locally determined ER status (either ER positive or negative).

Patients will be randomised to one of two treatment arms and will receive the following study treatments:

Arm A: Experimental Arm (n=82) Part I (Week 1-12) Epirubicin 90 mg/m2 by IV infusion on Day 1 every 21 days Cyclophosphamide 600 mg/m2 by IV infusion on Day 1 every 21 days Lapatinib 1000 mg orally once daily continuously Loperamide as required for the proactive management of diarrhoea (see Section 5.13.6)

Part II (Week 13-24) Paclitaxel 80 mg/m2 by IV infusion on Day 1 of each week Lapatinib 1000 mg orally once daily continuously Loperamide as required for the proactive management of diarrhoea (see Section 5.13.6)

Arm B: Reference Arm (n=82):

Part I (Week 1-12) Epirubicin 90 mg/m2 by IV infusion on Day 1 every 21 days Cyclophosphamide 600 mg/m2 by IV infusion on Day 1 every 21 days Part II (Week 13-24) Paclitaxel 80 mg/m2 by IV infusion on Day 1 of each week Trastuzumab 4 mg/kg IV load followed by 2 mg/kg IV Day 1 of each week

The primary study period includes the screening phase, administration of randomized neo-adjuvant study treatment, and assessments up to the primary endpoint assessment at the time of definitive breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent approved by an Independent Ethics Committee (IEC) and obtained prior to any study specific screening procedures.
2. Female patients aged ≥18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 -1.
4. Histologically confirmed, previously untreated, operable Stage I-IIIA invasive breast cancer:

   * Primary tumour greater than 1 cm in diameter measured by clinical examination and confirmed by at least one imaging study (mammography, breast ultrasound or MRI).
   * In the case of a multifocal tumour (defined as the presence of two or more foci of cancer within the same breast quadrant), the largest lesion must be >1 cm and is designated as the "target" lesion for all subsequent tumour evaluations.
5. Over expression and/or amplification of ErbB2 in the invasive component of the primary tumour according to one of the following definitions. Central laboratory confirmation is not required prior to randomization, but tumour samples must be available for banking and retrospective confirmation.

   • 3+ over expression by IHC (>30% of invasive tumour cells);
   * 2+ or 3+ (in 30% or less neoplastic cells) over expression by IHC AND in situ hybridization (FISH/CISH) test demonstrating ErbB2 gene amplification;
   * ErbB2 gene amplification by FISH/CISH (>6 ErbB2 gene copies per nucleus, or a FISH ratio [ErbB2 gene copies to chromosome 17 signals] of >2.2.) Patients with a negative or equivocal overall result (FISH test ratio of ≤2.2, ≤6.0 ErbB2 gene copies per nucleus) and staining scores of 0,1+, 2+ or 3+ (in 30% or less neoplastic cells) by IHC are NOT eligible for participation in the trial.
6. Known ER and PgR hormone receptor status.
7. LVEF within institutional normal range (evaluated by multiple-gated acquisition [MUGA] or echocardiography).
8. Women of childbearing potential must have a negative serum pregnancy test within 14 days (preferably 7 days) of first dose of study treatment and agree to use effective contraception, as defined in Section 7.3.2, during the study and for 28 days following the last dose of study drug.
9. Adequate baseline organ function defined by:

   • Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,

   • Hemoglobin ≥ 9 g/dL,

   • Platelet count ≥ 100 x 109/L,

   • Serum bilirubin ≤1.5 x ULN. In the case of known Gilbert´s syndrome, < 2x ULN is allowed,

   • ALT and AST ≤ 2.5 x ULN,

   • Alkaline phosphatase ≤ 2.5 x ULN,
   * Serum creatinine ≤ 1.6 mg/dL or calculated creatinine (Cockcroft and Gault ) clearance ≥50mL/m.
10. Patient agrees to make available tumour tissue samples for submission to the central laboratory for planned as well as future translational research.
11. French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

    -

Exclusion Criteria:

1. Metastatic, locally advanced, or inflammatory breast cancer as defined by the AJCC (7th Edition).
2. Bilateral breast cancer.
3. Multicentric breast cancer (defined as the presence of two or more foci of cancer in different quadrants of the same breast).
4. Any prior treatment for primary breast cancer (other than excision of tumour in the contralateral breast, and provided that the patient did not previously receive adjuvant radiotherapy or chemotherapy, all of which exclude the patient).
5. Concurrent participation in another clinical trial involving anti-cancer investigational drug or administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment.
6. History of any prior malignancy in previous 5 years (patients with a history of completely resected non-melanoma skin cancer or successfully treated carcinoma in situ of the cervix are eligible).
7. History of significant comorbidities that interfere with the conduct of the study, or evaluation of the results, or with informed consent.
8. Active infection.
9. Peptic ulcer or unstable diabetes mellitus within 8 weeks prior to study enrolment.
10. Clinically significant (i.e. active) cardiovascular disease, including cerebrovascular accident (≤6 months before enrolment), myocardial infarction (≤6 months before enrolment), unstable angina, New York Heart Association (NYHA) ≥ grade 2 congestive heart failure, serious cardiac arrhythmia requiring medication during the study and that might interfere with regularity of the study treatment, or not controlled by medication.
11. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
12. Lactating women.
13. Subjects unable to swallow and retain orally administered medication or with any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome, major resection of the stomach or bowels, or ulcerative colitis are also excluded.
14. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
15. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to any of the study drugs, active ingredients, or excipients that contraindicates their participation.
16. Concomitant use of CYP3A4 inhibitors or inducers.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) in the breast | At the time of definitive surgery

SECONDARY OUTCOMES:
pCR rate in the breast and axilla | At the time of definitive surgery
Overall response rate (complete plus partial response) in the breast and axilla according to RECIST 1.1 criteria | This will be measured at week 13 and post treatment prior to surgery
The breast conservation rate | At the time of definitive surgery

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- GSK Investigational Site, Graz, Austria
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gyula
- GSK Investigational Site, Oslo, Norway
- GSK Investigational Site, Castellon, Spain